CLINICAL TRIAL: NCT00459368
Title: Adherence Feedback for Improving Respiratory Medication Use
Brief Title: Using Information Technology to Improve Asthma Adherence
Acronym: AFFIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: L. Keoki Williams, MD, MPH, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL079055 (NIH)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-06

CONDITIONS: Asthma; Patient Compliance
Keywords: asthma; patient compliance; metered dose inhalers; corticosteroids; health behaviour; prevention & control
MeSH Terms: conditions — Asthma; Patient Compliance | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): In this cluster-randomized trial physicians practicing at intervention clinic sites will receive adherence information on their patients with asthma who are currently taking an inhaled corticosteroid medication. This information will be available to them via our electronic prescribing software to discuss with patients at the time of the visit. Physicians at these sites also receive standardized training in how to interpret and intervene when poor adherence is identified.
  Interventions: Behavioral: Feedback of patient adherence information
- II (Active Comparator): Physician practicing at control sites are given standard training in how to intervene on poor adherence, but no patient adherence information is provided to these clinicians via electronic prescribing software.
  Interventions: Behavioral: Active control group

INTERVENTIONS:
Behavioral: Feedback of patient adherence information — Patient inhaled corticosteroid adherence information is being provided to physicians at clinic sites randomized to the intervention arm. Adherence information is available via electronic prescribing software, and so is available to physicians when writing, renewing, or viewing medications. Physicians at intervention sites also receive standard training in how to interpret adherence metrics and how to intervene on poor adherence.
  Other Names: Adherence feedback
  Arms: I
Behavioral: Active control group — Physician practicing at control sites are given standard training in how to intervene on poor adherence, but no patient adherence information is provided to these clinicians via electronic prescribing software.
  Other Names: Standard care
  Arms: II

SUMMARY:
The purpose of this study is to determine whether providing patient medication adherence information on inhaled corticosteroid use to clinicians will result in improved patient adherence and asthma control.

DETAILED DESCRIPTION:
In 2001 an estimated 31.1 million people in the United States reported ever having had an asthma diagnosis. Asthma is a leading cause of preventable hospitalizations, and it accounts for an estimated 14 million days of missed school and 100 million days of restricted activity yearly.

The routine use of anti-inflammatory medications, particularly inhaled corticosteroids (ICS), in the treatment of asthma can markedly improve symptoms and reduce complications. Yet, evidence suggests that these medications are under-prescribed by physicians and poorly taken by patients. For example, in one study of asthma patients enrolled in a large, California HMO only 71.7% of patients with severe symptoms reported having a steroid inhaler, and only 53.6% of those reported using it daily in the preceding month. Using electronic monitoring devices to record inhaler use, researchers have estimated that patients use their ICS as directed 20 to 73% of the time. Using claims-based measures of adherence we have shown that adherence to inhaled steroids is inversely correlated with the frequency of oral steroid use and asthma-related emergency room visits. In addition, these measures suggest that non-adherence to ICS is an independent predictor of asthma-related hospitalizations. In our study population, we estimated that 60% of asthma-related hospitalizations were attributable to poor adherence to ICS. Together these findings suggest that increasing ICS use may improve asthma outcomes.

Studies employing health-behavioral models of adherence suggest that medication adherence is associated with treatment-related concerns regarding complications, efficacy, and benefits. Unfortunately, the results of behavioral and educational interventions to improve adherence have been disappointing. Despite, in some cases, considerable time spent with patients, these interventions have at best resulted in modest adherence improvements. Given the time, training, and resources required to implement these interventions, they are unlikely to be widely adopted in the clinical setting. Some recent studies, however, suggest that providing adherence data to clinicians may improve patient adherence. In one, clinicians gave repeated feedback to patients regarding ICS adherence; this resulted in sustained improvements over the study period. Unfortunately, this small study did not find differences in asthma outcomes.

In this proposal we seek to test an asthma adherence intervention specifically designed for use in the clinical setting. Adherence measures will be generated by linking currently available electronic data. In this cluster-randomized trial, primary care physician-practice groups will be randomized to receive asthma medication adherence information electronically for patients with asthma associated with these practices. In addition to ICS adherence information, clinicians in intervention practices will have data on patient beta-agonist use to better tailor ICS therapy to disease severity.

Eligible patients with asthma will be identified prior to randomizing practices and will be invited to participate. Patient surveys will be sent in the pre-intervention survey and in the post-intervention period. Patient-level outcomes will be assessed through the medical record, patient surveys, and claims data.

We will perform an intention-to-treat analysis with all eligible patients identified pre-randomization included in the analysis (the primary analysis). This study is powered to allow for only 60% of the eligible patient population being seen within the first 6-months (i.e., no effect in 40% of the patient population). As a secondary analysis, we will perform a modified intention-to-treat (or per protocol) analysis, whereby we will analyze the results of only those patients in both study arms seen within the first 6-months of the intervention.

ELIGIBILITY:
Inclusion Criteria (patient-level):

* Age 5-56 years
* Physician diagnosis of asthma
* Continuous HMO enrollment with prescription drug rider
* Electronic prescription of an inhaled corticosteroid

Exclusion Criteria (patient-level):

* Diagnosis of chronic obstructive pulmonary disease
* Diagnosis of congestive heart failure

Inclusion Criteria (practice-level):

* Primary care practice (i.e., pediatrics, family practice, or internal medicine) within the health system. A practice is defined as a group of physicians who by virtue of speciality or geography care for a relatively contained population of patients and who cross-cover the care of these patients.

Exclusion Criteria (practice-level):

* None

Ages: 5 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2698 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Keoki Williams, MD, MPH, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Self-reported asthma prevalence and control among adults--United States, 2001. MMWR Morb Mortal Wkly Rep. 2003 May 2;52(17):381-4. PMID 12765201
- [Background] Legorreta AP, Christian-Herman J, O'Connor RD, Hasan MM, Evans R, Leung KM. Compliance with national asthma management guidelines and specialty care: a health maintenance organization experience. Arch Intern Med. 1998 Mar 9;158(5):457-64. doi: 10.1001/archinte.158.5.457. PMID 9508223
- [Background] Cochrane MG, Bala MV, Downs KE, Mauskopf J, Ben-Joseph RH. Inhaled corticosteroids for asthma therapy: patient compliance, devices, and inhalation technique. Chest. 2000 Feb;117(2):542-50. doi: 10.1378/chest.117.2.542. PMID 10669701
- [Background] Williams LK, Pladevall M, Xi H, Peterson EL, Joseph C, Lafata JE, Ownby DR, Johnson CC. Relationship between adherence to inhaled corticosteroids and poor outcomes among adults with asthma. J Allergy Clin Immunol. 2004 Dec;114(6):1288-93. doi: 10.1016/j.jaci.2004.09.028. PMID 15577825
- [Background] Apter AJ, Boston RC, George M, Norfleet AL, Tenhave T, Coyne JC, Birck K, Reisine ST, Cucchiara AJ, Feldman HI. Modifiable barriers to adherence to inhaled steroids among adults with asthma: it's not just black and white. J Allergy Clin Immunol. 2003 Jun;111(6):1219-26. doi: 10.1067/mai.2003.1479. PMID 12789220
- [Background] Schmaling KB, Afari N, Blume AW. Assessment of psychological factors associated with adherence to medication regimens among adult patients with asthma. J Asthma. 2000 Jun;37(4):335-43. doi: 10.3109/02770900009055457. PMID 10883744
- [Background] Leickly FE, Wade SL, Crain E, Kruszon-Moran D, Wright EC, Evans R 3rd. Self-reported adherence, management behavior, and barriers to care after an emergency department visit by inner city children with asthma. Pediatrics. 1998 May;101(5):E8. doi: 10.1542/peds.101.5.e8. PMID 9565441
- [Background] Bender B, Milgrom H, Apter A. Adherence intervention research: what have we learned and what do we do next? J Allergy Clin Immunol. 2003 Sep;112(3):489-94. doi: 10.1016/s0091-6749(03)01718-4. PMID 13679805
- [Background] McDonald HP, Garg AX, Haynes RB. Interventions to enhance patient adherence to medication prescriptions: scientific review. JAMA. 2002 Dec 11;288(22):2868-79. doi: 10.1001/jama.288.22.2868. PMID 12472329
- [Background] Schectman JM, Schorling JB, Nadkarni MM, Voss JD. Can prescription refill feedback to physicians improve patient adherence? Am J Med Sci. 2004 Jan;327(1):19-24. doi: 10.1097/00000441-200401000-00005. PMID 14722392
- [Background] Onyirimba F, Apter A, Reisine S, Litt M, McCusker C, Connors M, ZuWallack R. Direct clinician-to-patient feedback discussion of inhaled steroid use: its effect on adherence. Ann Allergy Asthma Immunol. 2003 Apr;90(4):411-5. doi: 10.1016/S1081-1206(10)61825-X. PMID 12722963
- [Background] Donner A, Klar N. Pitfalls of and controversies in cluster randomization trials. Am J Public Health. 2004 Mar;94(3):416-22. doi: 10.2105/ajph.94.3.416. PMID 14998805
- [Background] Campbell MK, Elbourne DR, Altman DG; CONSORT group. CONSORT statement: extension to cluster randomised trials. BMJ. 2004 Mar 20;328(7441):702-8. doi: 10.1136/bmj.328.7441.702. No abstract available. PMID 15031246
- [Derived] Ahmedani BK, Peterson EL, Wells KE, Williams LK. Examining the relationship between depression and asthma exacerbations in a prospective follow-up study. Psychosom Med. 2013 Apr;75(3):305-10. doi: 10.1097/PSY.0b013e3182864ee3. Epub 2013 Feb 25. PMID 23440228
- [Derived] Ahmedani BK, Peterson EL, Wells KE, Rand CS, Williams LK. Asthma medication adherence: the role of God and other health locus of control factors. Ann Allergy Asthma Immunol. 2013 Feb;110(2):75-9.e2. doi: 10.1016/j.anai.2012.11.006. Epub 2012 Dec 7. PMID 23352524
- [Derived] Williams LK, Peterson EL, Wells K, Campbell J, Wang M, Chowdhry VK, Walsh M, Enberg R, Lanfear DE, Pladevall M. A cluster-randomized trial to provide clinicians inhaled corticosteroid adherence information for their patients with asthma. J Allergy Clin Immunol. 2010 Aug;126(2):225-31, 231.e1-4. doi: 10.1016/j.jaci.2010.03.034. Epub 2010 May 31. PMID 20569973
- [Derived] Paris J, Peterson EL, Wells K, Pladevall M, Burchard EG, Choudhry S, Lanfear DE, Williams LK. Relationship between recent short-acting beta-agonist use and subsequent asthma exacerbations. Ann Allergy Asthma Immunol. 2008 Nov;101(5):482-7. doi: 10.1016/S1081-1206(10)60286-4. PMID 19055201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Health system primary care providers (i.e., in the areas of family practice, internal medicine, and pediatrics) were invited to participate. Physicians who consented to participate were grouped according to practice.
Pre-assignment Details: One hundred ninety-two (92%) of the 207 primary care staff clinicians, representing 34 pre-defined primary care practices within the health system, agreed to participate. One clinic was not included a priori since it functioned as the primary resident clinic for internal medicine trainees.
Groups:
- Patient Medication Adherence Feedback: In this cluster-randomized trial physicians practicing at intervention clinic sites will receive adherence information on their patients with asthma who are currently taking an inhaled corticosteroid medication. This information will be available to them via our electronic prescribing software to discuss with patients at the time of the visit. Physicians at these sites also receive standardized training in how to interpret and intervene when poor adherence is identified.
- Usual Care: Physician practicing at control sites are given standard training in how to intervene on poor adherence, but no patient adherence information is provided to these clinicians via electronic prescribing software.
Period: Overall Study
Arm/Group | Patient Medication Adherence Feedback | Usual Care
Started | 1335 | 1363
Completed | 1040 | 1034
Not Completed | 295 | 329

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Medication Adherence Feedback | Usual Care | Total
Number analyzed (Participants) | 1335 | 1363 | 2698
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 591 | 604 | 1195
  Between 18 and 65 years | 744 | 759 | 1503
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.6 (37.3) | 27.7 (38.5) | 26.6 (37.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 737 | 753 | 1490
  Male | 598 | 610 | 1208
Region of Enrollment [Number; unit: participants]
  United States | 1335 | 1363 | 2698

OUTCOME MEASURES:

1. Primary Outcome: Patient Adherence to Inhaled Corticosteroids (ICS)
Description: Adherence to ICS medication was measured during the last 3 months of the intervention (i.e., for the time period of 9-12 months post-randomization). Adherence was measured using pharmacy claims data, and represents the percent of prescribed medication taken. The normal range for this value is 0-100%.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Percent of ICS medication taken
Arm/Group | Patient Medication Adherence Feedback | Usual Care
Number analyzed (Participants) | 1335 | 1363
Percent of ICS medication taken | 21.3 (2.5) | 23.3 (2.2)

2. Secondary Outcome: Asthma-related Emergency Room Visits
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Asthma-related Hospitalizations
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Oral Steroid Use
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Patient Self-efficacy to ICS Treatment
Time Frame: survey following intervention period
Reporting Status: Not Posted

6. Secondary Outcome: Readiness to Improve ICS Adherence (Transtheoretical Model)
Time Frame: survey following intervention period
Reporting Status: Not Posted

7. Secondary Outcome: Patient-physician Communication (Patient Reported Measure)
Time Frame: survey following intervention period
Reporting Status: Not Posted

8. Secondary Outcome: Patient Medical Care Costs
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Patient Medication Adherence Feedback | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/1335 | 0/1363
Other Adverse Events (participants affected / at risk) | 0/1335 | 0/1363

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No